CLINICAL TRIAL: NCT01812785
Title: Study to Investigate the Causes of Fever in Children Living in Urban Dar es Salaam and Rural Ifakara
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: Feverstudy; SNSF (Other Grant/Funding Number: SNSF grants # 3270B0-109696 and # IZ70Z0-124023)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Fever; Children; Infectious Diseases
Keywords: Fever; Children; Non-malaria fevers; Diagnosis
MeSH Terms: conditions — Fever; Communicable Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal is to improve the evidence-based management of fever cases seen in outpatient clinics in malaria endemic countries, through a better understanding of the value of accurate malaria diagnosis, and through an improved understanding of the other causes of fever in children. The objective is to describe systematically (as much as possible) the etiologies of fever in children in an urban and in a rural environment of sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* axillary temperature of 38°C or more
* first consultation for the present problem
* history of fever lasting for one week or less
* main complaint was not an injury or trauma
* no report of an antimalarial or antibiotic medicine taken during the previous week

Exclusion Criteria:

* severe malnutrition
* categorized as P1 (requiring immediate live saving procedures)

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive patients aged 2 months to 10 years presenting at the outpatient clinic of Amana district hospital in Dar es Salaam, and at the outpatient clinic of St-Francis designated-district hospital in Ifakara, Kilombero District.
Sampling Method: Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proportion of each disease and proportion of fevers of unknown origin in febrile children aged 2 months to 10 years attending an Outpatient Department of a district hospital in Dar es Salaam and in Ifakara | December 2011

SECONDARY OUTCOMES:
Clinical and laboratory predictors of each disease | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, prof, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- Tanzania (2):
  - Amana district hospital, Dar es Salaam, Dar es Salaam Region
  - St Francis hospital, Ifakara, Morogoro